CLINICAL TRIAL: NCT04108520
Title: Association of Diaphragmatic Exercises With the Functional Rehabilitation Protocol Effects on the Pulmonary Function of Individuals With Parkinson's Disease
Brief Title: Diaphragmatic Exercise on Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Director of Human Movement Department, Universidade Metodista de Piracicaba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25092019
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Exercises on respiratory muscle, 3 times per week, 1 hour peer day
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise with respiratory training

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease in the world, considering the central nervous system disorders that affect movement. In addition to motor impairment, the literature reinforces changes in ventilatory parameters, such as restrictive lung dysfunction, obstructive airway disease, and upper airway obstruction. Pulmonary disorders are more evident in patients in later and advanced stages of PD, and are responsible for most of the morbimortalities resulting from the disease. Objectives: To evaluate the effects of a protocol of diaphragmatic awareness, in association with the global exercises, on the pulmonary function of individuals with Parkinson's disease. Methods: This is an experimental, uncontrolled clinical trial. Participants are patients with Parkinson's disease referred for care at the UEAFTO / CER-II UEPA neurofunctional outpatient clinic whose records will be consulted for the collection of epidemiological data and postural assessment of cognitive functions through protocol Montreal Cognitive Assessment (Brazilian experimental version) and classification by modified Hoehn and Yahr scale. Those who meet the inclusion criteria will be evaluated through the evaluation form, Pulmonary Functional Status and Dyspnea Questionnair protocol, submitted to Pulmonary Function Test and respiratory muscle strength assessment by Spirometry and Manovacuometry, respectively. They will be submitted to an intervention protocol prepared by the physiotherapy team of UEPA's Elderly Care Center for 20 sessions lasting 60 minutes twice a week, consisting of global exercises and diaphragmatic awareness, being re-evaluated in the 10th and 20th sessions. The protocol used will be registered in the Clinical Trials database. All participants will sign a Free and Informed Consent Form and the research will be submitted to analysis by the Human Research Ethics Committee of the University of the State of Pará (UEPA). The data collected will be tabulated in a Microsoft Excel 2016® worksheet for further statistical analysis using BioEstat® 5.3 software. Expected results: obtain an improvement in the variables related to pulmonary function in the experimental group after the application of the intervention protocol and in relation to the control group.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disease in the world, considering the central nervous system disorders that affect movement. In addition to motor impairment, the literature reinforces changes in ventilatory parameters, such as restrictive lung dysfunction, obstructive airway disease, and upper airway obstruction. Pulmonary disorders are more evident in patients in later and advanced stages of PD, and are responsible for most of the morbimortalities resulting from the disease. Objectives: To evaluate the effects of a protocol of diaphragmatic awareness, in association with the global exercises, on the pulmonary function of individuals with Parkinson's disease. Methods: This is an experimental, uncontrolled clinical trial. Participants are patients with Parkinson's disease referred for care at the UEAFTO / CER-II UEPA neurofunctional outpatient clinic whose records will be consulted for the collection of epidemiological data and postural assessment of cognitive functions through protocol Montreal Cognitive Assessment (Brazilian experimental version) and classification by modified Hoehn and Yahr scale. Those who meet the inclusion criteria will be evaluated through the evaluation form, Pulmonary Functional Status and Dyspnea Questionnair protocol, submitted to Pulmonary Function Test and respiratory muscle strength assessment by Spirometry and Manovacuometry, respectively. They will be submitted to an intervention protocol prepared by the physiotherapy team of UEPA's Elderly Care Center for 20 sessions lasting 60 minutes twice a week, consisting of global exercises and diaphragmatic awareness, being re-evaluated in the 10th and 20th sessions. The protocol used will be registered in the Clinical Trials database. All participants will sign a Free and Informed Consent Form and the research will be submitted to analysis by the Human Research Ethics Committee of the University of the State of Pará (UEPA). The data collected will be tabulated in a Microsoft Excel 2016® worksheet for further statistical analysis using BioEstat® 5.3 software. Expected results: to obtain an improvement in the variables related to pulmonary function in the experimental group after the application of the intervention protocol and in relation to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's of both genders
* No reports of respiratory diseases and / or other previous neurological complications in the assessment form
* Residents in the metropolitan area of Belém.

Exclusion Criteria:

* Patients with cognitive impairment or dementia
* Patients with previous respiratory conditions or another neurological condition.
* Patients with two consecutive absences or four absences alternating with treatment.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | post treatment in 3 days
  A digital manovacuometer will be used to measure respiratory muscle strength, providing maximum inspiratory pressure and Maximum Expiratory Pressure. A nasal clip will be used throughout the procedure to avoid air leakage. Thus, in order to obtain the measures of MIP, the volunteer is instructed to perform a maximal expiration and soon afterwards, through vocal encouragement, the individual will perform a maximum and sustained inspiratory effort for at least 2 seconds. Also, for the values of MEP, where the participant will perform a maximum inspiration before the maximum sustained respiratory effort. The PImax and PEmax maneuvers will first be learned, being executed 3 times by each member, adopting the values consistent with each other, with a difference of 10% between each result.

CONTACTS AND LOCATIONS:
Overall Officials: Lorena ZAHLUTH, phd, Study Chair — Universidade do Estado do Pará
Locations (1):
- Universidade do Estado do Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No